CLINICAL TRIAL: NCT03099330
Title: Phase I Study of Tolerance and Pharmacokinetics of TQ-B3139 in Patients With Advanced Cancer
Brief Title: A Phase I Study of TQ-B3139 on Tolerance and Pharmacokinetics
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQ-B3139-I-0001
Record Dates: First submitted 2017-03-28; First posted 2017-04-04 (Actual); Last update posted 2017-09-18 (Actual); Status verified 2017-03

CONDITIONS: Advanced Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- TQ-B3139 (Experimental): TQ-B3139 p.o. qd
  Interventions: Drug: TQ-B3139

INTERVENTIONS:
Drug: TQ-B3139 — TQ-B3139 p.o. qd

SUMMARY:
A study of TQ-B3139, inhibitor of ALK/C-Met tyrosine kinase, in patient with advanced cancer

DETAILED DESCRIPTION:
phase I of safety, pharmacokinetic and pharmacodynamic study of TQ-B3139. To recommend a reasonable dose and indication for subsequent research.

ELIGIBILITY:
Inclusion Criteria:

* Histological documentation of Advanced solid tumors
* Lack of the standard treatment or treatment failure
* 18-65years,ECOG PS:0-1,Life expectancy of more than 3 months
* Patients with anti-treatment or surgery within 4 weeks
* Main organs function is normal
* Women of childbearing potential should agree to use and utilize an adequate method of contraception (such as intrauterine device，contraceptive and condom) throughout treatment and for at least 6 months after study is stopped；the result of serum or urine pregnancy test should be negative within 7 days prior to study enrollment，and the patients required to be non-lactating；Man participants should agree to use and utilize an adequate method of contraception throughout treatment and for at least 6 months after study is stopped
* Patients should participate in the study voluntarily and sign informed consent

Exclusion Criteria:

* Patients participated in other anticancer drug clinical trials within 4 weeks
* Blood pressure unable to be controlled(systolic pressure>140 mmHg，diastolic pressure>90 mmHg).

Patients with Grade 1 or higher myocardial ischemia, myocardial infarction or malignant arrhythmias(including QT≥470ms)

* Patients with non-healing wounds or fractures
* Patients with drug abuse history and unable to get rid of or Patients with mental disorders
* History of immunodeficiency
* Patients with concomitant diseases which could seriously endanger their own safety or could affect completion of the study according to investigators' judgment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-07-19 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
The maximum tolerated dose (MTD) of TQ-B3139 | 48 weeks
  The highest dose at which no more than 33% of the subjects experience a dose-limiting toxicity (DLT) during treatment
The type of dose-limiting toxicity(ies) (DLT[s]) of TQ-B3139 | For 4 weeks for DLTs
  Subjects within 28 days after treatment appear the following toxicity reaction relate to the drug ：III °or above of non-hematological toxicity,IV°hematological toxicity ,Neutropenia associated with fever
Pharmacokinetics of TQ-B3139 (in whole blood):Peak Plasma Concentration(Cmax) | up to 28 Days (endpoint when the two consecutive time points of blood drug concentration <150 DPM/mL)
  Peak Plasma Concentration(Cmax),Cmax in ng/mL.In the study of single-dose, full PK profiles will be obtained at H0/H1/H2/H3/H4/H6/H10/H24/H34/H48/H72/H96/H120/H144（H means Hour）.In the study of multiple-dose,full PK profiles will be obtained at D1/D4/D8/D15/D21/D28（D means Day）.
Pharmacokinetics of TQ-B3139 (in whole blood):Peak time（Tmax） | up to 28 Days (endpoint when the two consecutive time points of blood drug concentration <150 DPM/mL)
  Peak time（Tmax）,Tmax in h.In the study of single-dose, full PK profiles will be obtained at H0/H1/H2/H3/H4/H6/H10/H24/H34/H48/H72/H96/H120/H144（H means Hour）.In the study of multiple-dose,full PK profiles will be obtained at D1/D4/D8/D15/D21/D28（D means Day）.
Pharmacokinetics of TQ-B3139 (in whole blood):Half life（t1/2） | up to 28 Days (endpoint when the two consecutive time points of blood drug concentration <150 DPM/mL)
  Half life（t1/2）,t1/2 in h.In the study of single-dose, full PK profiles will be obtained at H0/H1/H2/H3/H4/H6/H10/H24/H34/H48/H72/H96/H120/H144（H means Hour）.In the study of multiple-dose,full PK profiles will be obtained at D1/D4/D8/D15/D21/D28（D means Day）.
Pharmacokinetics of TQ-B3139 (in whole blood):Area under the plasma concentration versus time curve (AUC) | up to 28 Days (endpoint when the two consecutive time points of blood drug concentration <150 DPM/mL)
  Area under the plasma concentration versus time curve (AUC), AUC in ng.h/mL.In the study of single-dose, full PK profiles will be obtained at H0/H1/H2/H3/H4/H6/H10/H24/H34/H48/H72/H96/H120/H144（H means Hour）.In the study of multiple-dose,full PK profiles will be obtained at D1/D4/D8/D15/D21/D28（D means Day）.
Pharmacokinetics of TQ-B3139 (in whole blood):Clearance（CL） | up to 28 Days (endpoint when the two consecutive time points of blood drug concentration <150 DPM/mL)
  Clearance（CL）,CL in L/h.In the study of single-dose, full PK profiles will be obtained at H0/H1/H2/H3/H4/H6/H10/H24/H34/H48/H72/H96/H120/H144（H means Hour）.In the study of multiple-dose,full PK profiles will be obtained at D1/D4/D8/D15/D21/D28（D means Day）.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | each 28 days up to intolerance the toxicity or PD (up to 24 months)

CONTACTS AND LOCATIONS:
Locations (1):
- Sun-Yat-Sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ma Y, Zhao H, Xue J, Liu L, Yang N, Zhang Y, Yang H, Hong S, Xiong Y, Zhang Z, Zeng L, Pan H, Zhou C, Zhang Y, Wang X, Han X, Wan X, Shao Y, Liu J, Yang Y, Huang Y, Zhao Y, Fang W, Li S, Zhang L. First-in-human phase I study of TQ-B3139 (CT-711) in advanced non-small cell lung cancer patients with ALK and ROS1 rearrangements. Eur J Cancer. 2022 Sep;173:238-249. doi: 10.1016/j.ejca.2022.06.037. Epub 2022 Aug 5. PMID 35940055